CLINICAL TRIAL: NCT01274624
Title: A Multicenter Phase 1 Study of Intravenous Administration of REOLYSIN® (Reovirus Type 3 Dearing) in Combination With Irinotecan/Fluorouracil/Leucovorin (FOLFIRI) and Bevacizumab in FOLFIRI Naive Patients With KRAS Mutant Metastatic Colorectal Cancer
Brief Title: Study of REOLYSIN® in Combination With FOLFIRI and Bevacizumab in FOLFIRI Naive Patients With KRAS Mutant Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 022
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: KRAS Mutant Metastatic Colorectal Cancer
Keywords: Colorectal; Cancer; REOLYSIN®; Chemotherapy; FOLFIRI; Reovirus; Oncolytic virus; Fluorouracil; Irinotecan; Leucovorin; Bevacizumab
MeSH Terms: conditions — Neoplasms | interventions — reolysin; Irinotecan; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN® — 1 hour intravenous infusion administered on Days 1, 2, 3, 4, and 5 every 4 weeks.
  Other Names: Reovirus serotype 3 Dearing Strain
Drug: Irinotecan — 90-minute intravenous infusion on Day 1 every 2 weeks. Dose levels of 125 mg/m2, 150 mg/m2, 150 mg/m2, 180 mg/m2.
Drug: Leucovorin — 2-hour infusion of 400 mg/m2 on Day 1 every 2 weeks.
Drug: Fluorouracil (5-FU) — 400 mg/m2 intravenous bolus followed by 2400 mg/m2 as a continuous intravenous infusion over 46 hours administered on Day 1 every 2 weeks.
Drug: Bevacizumab — 30, 60 or 90 minute infusion on Day 1 every 2 weeks. Dose level 5 mg/kg.

SUMMARY:
This is a Phase 1 dose-escalation study with three dose levels to determine the maximum tolerated dose of REOLYSIN® combined with FOLFIRI and bevacizumab.

DETAILED DESCRIPTION:
Reovirus Serotype 3 - Dearing Strain (REOLYSIN®) is a naturally occurring, ubiquitous, non-enveloped human reovirus. Reovirus has been shown to replicate selectively in Ras-transformed cells causing cell lysis. Activating mutations in ras or mutation in oncogenes signaling through the ras pathway may occur in as many as 80% of human tumors. The specificity of the reovirus for Ras-transformed cells, coupled with its relatively nonpathogenic nature in humans, makes it an attractive anti-cancer therapy candidate. Eligible patients for this study include those with histologically confirmed cancer of the colon or rectum with Kras mutation and measurable disease.

Cetuximab and panitumumab have shown to be ineffective in patients whose tumors have a KRAS mutation. Therefore, currently, for patients with a KRAS mutation, the only option after failure of front-line therapy is irinotecan or FOLFIRI. Over the past year, two randomized phase III trials have demonstrated that OS and PFS for these patients increase when bevacizumab is combined with the standard FOLFIRI therapy.

The trial is a Phase I dose escalation study with four dose levels, comprising cohorts of three to six patients, to determine a maximum tolerated dose and dose-limiting toxicities with the combination of REOLYSIN®, bevacizumab, and FOLFIRI. FOLFIRI and bevacizumab will be administered on the first day of a two week (14-day) cycle, while REOLYSIN® will be administered on days one through five of a four week (28-day) cycle.

The study is expected to enroll 20 to 32 patients.

ELIGIBILITY:
Inclusion Criteria: Each patient MUST:

* Have histologically confirmed cancer of the colon or rectum with radiologically documented and measurable metastases (high CEA alone is insufficient for study entry).
* Have received an oxaliplatin-based chemotherapy regimen in the metastatic setting or relapsed within 6 months of completion of adjuvant therapy containing oxaliplatin.
* Not have received prior FOLFIRI or irinotecan in the metastatic setting.
* Have his/her tumor assessed for KRAS status and found to be mutation positive.
* Have NO continuing acute toxic effects (except alopecia) of any prior radiotherapy, chemotherapy, or surgical procedures, i.e., all such effects must have been resolved.
* Be at least 18 years of age.
* Have an ECOG Performance Score of ≤ 2.
* Have a life expectancy of at least 3 months.
* Have baseline laboratory results as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9 [SI unit 10^9/L]
  * Platelets ≥ 100 x10^9 [SI units 10^9/L] (without platelet transfusion)
  * Hemoglobin ≥ 9.0 g/dL [SI units gm/L] (with or without RBC transfusion)
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Bilirubin ≤ ULN
  * AST/ALT ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
  * Negative pregnancy test for females with childbearing potential.
  * Proteinuria < grade 2.
* Have signed an informed consent indicating that the patient is aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
* Be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.
* Be medically eligible to receive bevacizumab

Exclusion Criteria: No patient may:

* Receive concurrent therapy with any other investigational anticancer agent while on study.
* Have previously received irinotecan or FOLFIRI in the metastatic setting (patient is eligible if he/she had received irinotecan or FOLFIRI as adjuvant therapy more than 6 months before entry into the study)
* Have brain metastases.
* Be on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Have received >20 Gy of radiation to the pelvis.
* Have received chemotherapy, immunotherapy, hormonal therapy or had major surgery within 28 days; or received radiotherapy within 14 days; or minor surgery within 7 days prior to receiving the study drug.
* Be a pregnant or breast-feeding woman. Female patients of childbearing potential must agree to use effective contraception, be surgically sterile, or be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. Barrier methods are a recommended form of contraception.
* Have clinically significant cardiac disease (New York Heart Association, Class III or IV) including pre-existing arrhythmia, uncontrolled angina pectoris, myocardial infarction within 1 year prior to study entry, or Grade 2 or higher compromised left ventricular ejection fraction.
* Have dementia or altered mental status that would prohibit informed consent.
* Have any other acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.
* Have uncontrolled hypertension, proteinuria, or recent major surgery (all clinical parameters related to bevacizumab use). Any other clinical parameter considered important should be discussed with the medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2018-02 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity to define maximum tolerated dose and recommended Phase 2 dose | During the first cycle of treatment (4 week cycle)
Pharmacokinetic parameters for irinotecan and 5-FU when combined with REOLYSIN® | During the first cycle of treatment (4 week cycle)

SECONDARY OUTCOMES:
CEA and Objective Response, Clinical Benefit Rate (PR, CR, SD), progression-free survival, and overall survival (PFS and OS) | Assessed every 8 weeks until disease progression or death
Safety and tolerability of REOLYSIN® when administered in combination with FOLFIRI and bevacizumab | During study and within 30 days of the last dose of REOLYSIN
Correlative studies including determination of specific genetic mutations and aberrant signalling pathways from tumor tissue to identify novel biomarkers of response and efficacy | During and within 30 days of the last dose of REOLYSIN®
In vitro studies in human-derived colorectal cancer cells including the isogenic cell lines, to study the mechanism and scientific basis of synergy between irinotecan and reovirus | During study and within 30 days of the last dose of REOLYSIN®

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York Presbyterian Hospital/ Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York